CLINICAL TRIAL: NCT03561324
Title: Intraoperative Imaging of a PET Positive Lymph Node(s) Using 18FDG and a Dual-Mode, Hand-Held Intraoperative Imager
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI leaving institution/no funding
Sponsor: University of Arkansas (Other)
Collaborators: Radiation Monitoring Devices, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 217729
Record Dates: First submitted 2018-05-31; First posted 2018-06-19 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Head and Neck Neoplasms
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Use of IntraOperative Imaging Probe (Experimental): The sterilized (Imaging Beta Probe) IBP will be used intraoperatively in surgical wounds for localization of tumor sites and detecting completeness of excision vs. positive margins.
  Interventions: Device: Imaging Beta Probe (IBP)

INTERVENTIONS:
Device: Imaging Beta Probe (IBP) — Using IBP for imaging of PET positive lymph nodes

SUMMARY:
This study is a prospective collection of data utilizing the Imaging Beta Probe (IBP) in patients with positron emission tomography (PET) positive disease. A pilot clinical study involving 5 patients will be conducted using the IBP. The sterilized IBP will be used intraoperatively in surgical wounds for localization of tumor sites and detecting completeness of excision vs. positive margins. The outcome of each of these studies will be documented and used to demonstrate clinical benefits of the new probe. The investigators will correlate the images from the probe of the Fludeoxyglucose (18FDG) positive tissue, both in-vivo and ex-vivo after dissection, with the previously performed PET scan and with the routine pathology results obtained on the surgical specimens.The experimental imaging modality studied in this protocol will be compared to clinically utilized modalities of ultrasound and PET/ CT. Localization between imaging modalities will be compared with respect to: detection and side of localization.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, 18- to 90-years old.
* Positive for PET positive disease in the neck.

Exclusion Criteria:

* Pregnant women (all women of child bearing potential will have undergone pregnancy testing as standard of care)
* Nursing or lactating women

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-06-20 (Actual); Primary Completion 2020-01-22 (Actual); Study Completion 2020-01-22 (Actual)

PRIMARY OUTCOMES:
Detection of PET positive disease | Day 1
  Localization between imaging modalities will be compared with respect to: detection (y/n) and side of localization (r/l).

CONTACTS AND LOCATIONS:
Overall Officials: Deanne L King, MD, Study Director — 501-686-5140
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No